CLINICAL TRIAL: NCT00981357
Title: A Phase 2a Randomized, Double-blinded, Double Dummy, Placebo And Active Controlled, Two-way Cross-over, Flare-enriched Multi-centre Clinical Trial To Examine The Pain Relief Produced By 2 Weeks Of Daily Oral Administration Of A Fatty Acid Amide Hydrolase (Faah) Inhibitor Pf-04457845 In Patients With Osteoarthritis Of The Knee.
Brief Title: A Study To Investigate Whether PF-04457845 Is Effective In Treating Pain, Is Safe And Tolerable In Patients With Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0541004; 2009-014734-16 (EudraCT Number)
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Cross-over evaluate the efficacy of PF-04457845 in relieving pain due to osteoarthritis OA knee osteoarthritis of knee pain due to osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04457845 followed by placebo (Experimental)
  Interventions: Drug: PF-04457845
- Placebo followed by PF-04457845 (Experimental)
  Interventions: Drug: PF-04457845
- Naproxen followed by placebo (Active Comparator)
  Interventions: Drug: Naproxen
- Placebo followed by Naproxen (Active Comparator)
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: PF-04457845 — PF-04457845 4 mg tablet once daily / matched placebo
  Arms: PF-04457845 followed by placebo
Drug: PF-04457845 — PF-04457845 4 mg tablet once daily / matched placebo
  Arms: Placebo followed by PF-04457845
Drug: Naproxen — Naproxen 500 mg tablet twice daily / matched placebo
  Arms: Naproxen followed by placebo
Drug: Naproxen — Naproxen 500 mg tablet twice daily / matched placebo
  Arms: Placebo followed by Naproxen

SUMMARY:
Inactivation of the FAAH (Fatty Acid Amide Hydrolase) enzyme has been shown to relieve pain and inflammation in animal studies. PF-04457845 has been shown to inactivate the FAAH enzyme in animals and healthy human volunteers. The purpose of this study is to evaluate whether PF-04457845 can inactivate the FAAH enzyme in patients experiencing pain due to OA and whether this results in these patients experiencing less pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of Osteoarthritis (OA) of the knee confirmed by X-ray
* Subjects must be willing and able to stop all current pain therapy for the duration of study. (Limited and specific pain therapy will be available throughout the study)
* Subjects can be male or female between the ages of 18 and 75 years inclusive, but female subjects must not be able become pregnant

Exclusion Criteria:

* Subjects must not have any condition or medical history that might interfere with their ability to complete the study assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of PF-04457845 (administered QD) versus placebo in relieving pain as measured by the WOMAC Pain sub-score in patients with osteoarthritis of the knee | 8 weeks
To evaluate the safety and tolerability of PF-04457845 in patients with osteoarthritis. | 10 weeks

SECONDARY OUTCOMES:
Efficacy of PF-04457845 (administered QD) versus placebo as measured by the WOMAC Stiffness domain score (Likert scale for 2 items, overall score ranges from 0-8) in patients with osteoarthritis of the knee. | 8 weeks
Efficacy of PF-04457845 (administered QD) versus placebo as measured by the WOMAC Physical Function domain score (Likert scale for 17 items, overall score ranges from 0-68) in patients with osteoarthritis of the knee. | 8 weeks
Efficacy of PF-04457845 (administered QD) versus placebo as measured by the WOMAC Total Score in patients with osteoarthritis of the knee. | 8 weeks
Efficacy of PF-04457845 (administered QD) versus placebo as measured by the Importance weighted Total WOMAC score in patients with osteoarthritis of the knee. | 8 weeks
Efficacy of PF-04457845 (administered QD) versus placebo as measured by the Daily pain diary over weeks 1 and 2 of each treatment period using an 11-point Numeric Rating Scale (NRS) in patients with osteoarthritis of the knee. | 8 weeks
Efficacy of PF-04457845 (administered QD) versus placebo as measured by the Subjects' use of rescue medication on either treatment. | 8 weeks
Summary of plasma concentrations of PF-04457845. | 8 weeks
Residual FAAH activity in leukocytes for subjects recruited prior to the interim analysis. | 8 weeks
Plasma fatty acid amide levels (OEA, PEA, LEA and AEA) for subjects recruited prior to the interim analysis. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (4):
  - Arthritis & Rheumatic Care Center, Miami, Florida
  - Miami Research Associates, Miami, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - CEDRA Clinical Research, LLC, San Antonio, Texas
- Diex Research Inc., Sherbrooke, Quebec, Canada
- Centrum for klinisk provning, Gothenburg, Sweden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0541004&StudyName=A%20Study%20To%20Investigate%20Whether%20PF-04457845%20Is%20Effective%20In%20Treating%20Pain%2C%20Is%20Safe%20And%20Tolerable%20In%20Patients%20With%20Osteoarthritis%20Of%20T